CLINICAL TRIAL: NCT00613184
Title: Comparison of Nylon Flocked Swabs and Saline Aspirates for Detection Respiratory Viruses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kern Medical Center (Other)
Collaborators: Medical Diagnostic Laboratories, LLC (Industry); Copan Innovation Murrietta, CA (Unknown)
Responsible Party: Paul Walsh MB BCh FACEP, Department of Emergency Medicine, Kern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: kmc06037
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Respiratory Syncytial Virus; Human Metapneumovirus; Influenza; Bronchiolitis; Pediatric
Keywords: Respiratory Syncytial virus; Bronchiolitis; Pediatric
MeSH Terms: conditions — Influenza, Human; Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Nylon Flocked swab Left Nasal Wash right
  Interventions: Device: Nylon Flocked swab (Nasal secretion sampling)
- 2 (Experimental): Nylon Flocked swab R Nasal Wash L
  Interventions: Device: Nylon Flocked swab (Nasal secretion sampling)
- 3 (Experimental): Nasal Wash Left Nylon Flocked swab Right
  Interventions: Device: Nylon Flocked swab (Nasal secretion sampling)
- 4 (Experimental): Nasal Wash R Nylon flocked swab L
  Interventions: Device: Nylon Flocked swab (Nasal secretion sampling)

INTERVENTIONS:
Device: Nylon Flocked swab (Nasal secretion sampling) — Nasal Aspirate Nylon Flocked swab
Device: Nylon Flocked swab (Nasal secretion sampling) — Nylon flocked swab Nasal Wash
  Arms: 1

SUMMARY:
Collection of nasal secretions from infants and toddlers for viral testing is usually done using the nasal washing technique described by Hall in 1975. This is cumbersome. Previous attempts to use swabs have been unsuccessful because the swabs didn't work well. A newly designed swab may work better and in this study we compare the new swab with the old style nasal washing.

.

DETAILED DESCRIPTION:
Collection of nasal secretions from infants and toddlers for viral testing is typically performed using the nasal saline aspirate technique described by Hall in 1975.

Nylon flocked swabs (NFS) and universal transport medium for room temperature (UTM-RT) (Copan Medical, Murrieta, CA) storage media have been found to be an effective collection and transport method for bacteria causing sexually transmitted infections.

We adapted these swabs and storage medium to collect respiratory viruses from children less than18 months old and compared detection rates using NFS and traditional nasal aspirates. We will determine the relative roles of the UTM-RT and NFS release and therefore measured viral detection rates of common respiratory pathogens in traditional saline aspirates stored in UTM-RT.

Our primary hypothesis is that nasal secretions collection using NFS stored in UTM-RT will lead to a higher detection rate of the respiratory viruses we arestudying; namely RSV, Influenza and human metapneumovirus from than collection of unpreserved saline nasal aspirates in children less than 18 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Treating clinican ordered RSV antigen testing

Exclusion Criteria:

* Refusal of consent
* Age > 18 months

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Viral detection rate by PCR | 0 not applicable

CONTACTS AND LOCATIONS:
Overall Officials: Paul Walsh, MD, Principal Investigator — Kern Medical Center & David Geffen School of Medicine UCLA